CLINICAL TRIAL: NCT02800837
Title: Multicenter Prospective Clinical Study of the STENTYS Xposition S for Treatment of Unprotected Left Main Coronary Artery Disease
Brief Title: Clinical Study to Evaluate the STENTYS Xposition S for Treatment of Unprotected Left Main Coronary Artery Disease
Acronym: TRUNC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Stentys (Industry)
Responsible Party: Sponsor
Other Study IDs: ST2016-01
Record Dates: First submitted 2016-05-09; First posted 2016-06-15 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-05

CONDITIONS: Coronary Artery Disease (Left Main)
Keywords: left main; stent; self-expandable; DES; Stentys
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Prospective, non-randomized, multi-center study assessing the long term safety and efficacy of the self expandable sirolimus eluting Xposition S stent in the treatment of unprotected left main coronary artery disease.

DETAILED DESCRIPTION:
In the treatment of unprotected left main coronary artery (ULMCA) disease, previous mono-center studies have shown promising results with the previous generation of the self-expandable STENTYS stent (paclitaxel eluting stent, delivered via withdrawal of a sheath).

The TRUNC study aims at assessing at large scale the Xposition S in the treatment of ULMCA disease. The Xposition S is a sirolimus eluting stent, mounted on a balloon delivery system. The study aims at collecting clinical practice routine data from 200 patients.

ELIGIBILITY:
Main Inclusion Criteria:

* Subject ≥ 18 years old;
* Presence of coronary artery stenosis in the unprotected Left Main (LM) Coronary Artery which is indicated for PCI and Xposition S stent treatment
* Left Main Coronary Artery reference vessel diameter ranging from 2.5 mm to 6.0 mm;
* The subject is able to provide voluntary informed consent, willing to comply with all study requirements and sign the written informed consent.

Main Exclusion Criteria:

* Recent STEMI (<1 month) ;
* SYNTAX score ≥ 33 ;
* Highly calcified lesions or excessive tortuosity at target lesion site;
* Subject unable to comply with dual antiplatelet therapy as recommended per guidelines;
* Planned cardiac surgery or valve intervention within the next 12 months.
* Participation to other investigational drug or device studies that have not reached their primary endpoint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery stenosis (unprotected left main coronary artery), indicated for Percutaneous Coronary Intervention (PCI) and Xposition S stent treatment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Clinical Endpoint- Target Lesion Failure (TLF) | 12 months post-procedure
  TLF defined as cardiac death, MI not attributable to a non target vessel, or clinically driven target lesion revascularization
Efficacy Endpoint - Angiographic Success | 12 months post-procedure
  Achievement of <20% final residual stenosis at target lesion (visual estimation) with TIMI 3 flow in main branch

SECONDARY OUTCOMES:
Procedural Success | 48 hours post procedure (hospital discharge)
  Angiographic success without occurence of death, target lesion related MI or target lesion revascularization prior to hospital discharge visit
TLF | 30 days post procedure
  TLF defined as cardiac death, Myocardial Infarction(MI) not attributable to a non target vessel, or clinically driven target lesion revascularization
Cardiac Death Rate | 30 days, 12 months and 24 months post procedure
MI rate (not attributable to a non target vessel) | 30 days, 12 months and 24 months post procedure
Clinically Driven Target Lesion Revascularization | 30 days, 12 months and 24 months post procedure
Stroke Events Rate | 30 days, 12 and 24 months post procedure
Stent Thrombosis Events Rate | 30-day, 12-month and 2 year post-procedure
Index Procedure Duration | End of the index procedure
Fluoroscopy Time, during Index Procedure | End of the index procedure
Acute Stent Malappositon by IVUS (IVUS Substudy) | End of the index procedure
  Assessed in a subset of patients
Minimal Lumen Area by IVUS (IVUS substudy) | End of the index procedure
  Assessed in a subset of patients

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (2):
  - Ferraroto Hospital - Catania University, Catania
  - Clinica Mediterranea, Naples
- St Gallen Kantonsspital, Sankt Gallen, Switzerland
- Bristol Heart Institute, Bristol, United Kingdom

REFERENCES:
- [Background] Briguori C, Visconti G, Donahue M, Focaccio A, Mitomo S, Kawamoto H, Nakamura S. The STENTYS(R) paclitaxel-eluting stent in the treatment of unprotected distal left main. Catheter Cardiovasc Interv. 2015 Sep;86(3):E131-9. doi: 10.1002/ccd.25874. Epub 2015 Feb 25. PMID 25639945